CLINICAL TRIAL: NCT06792981
Title: Effectiveness and Cost-effectiveness of an Online School-based Program for Reducing Risk Factors in Pre-adolescents (PRETA): Protocol for a Cluster Randomized Controlled Trial
Brief Title: Evaluation of a Digital School-Based Intervention for the Primary Prevention of Eating Disorders in Pre-Adolescents (PRETA Program)
Acronym: PRETA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: University of La Laguna (Other); Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other)
Responsible Party: Principal Investigator, Yolanda Ramallo Fariña, Coordinator of the Research Methodology and Data Analysis Group, Servicio Canario de Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIFIISC21/06
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Eating Disorders in Adolescence; Food Addiction
Keywords: eating disorders; school-based intervention; efficacy; efficiency; Universal Prevention Program; Online Health
MeSH Terms: conditions — Food Addiction; Feeding and Eating Disorders

STUDY DESIGN:
Masking Description: Data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will complete a baseline assessment and receive project information. Then, students from the schools randomly allocated to the intervention group will participate in the PRETA program, specifically designed for the primary prevention of Eating Disorders (ED) in a school setting. These sessions will involve educational activities and participatory dynamics to foster a healthy relationship with body image and eating. At the end of the program, participants will complete questionnaires to assess the outcomes.
  Additionally, parents and teachers in the intervention group will receive targeted training and resources.
  Interventions: Other: Universal primary prevention program based on ICTs
- Control Group (No Intervention): The students randomly allocated to control condition will not receive any type of intervention. They will continue with their regular school activities but will complete the questionnaires and surveys to contrast the effects of the intervention.

INTERVENTIONS:
Other: Universal primary prevention program based on ICTs — The intervention adopts a multicomponent approach, addressing three agents in the prevention and management of eating disorders: parents, teachers and students.
  1. Intervention with parents:
     Parents will receive specific materials, including an informative guide on early identification of warning signs, promoting healthy lifestyle habits, and fostering effective communication with their children.
  2. Intervention with teachers:
     A two-hour in-person session will train teachers on platform use and provide tools for eating disorder prevention through role-playing techniques. Online resources will complement the training, while researchers ensure adherence via weekly follow-ups and parent reminders.
  3. e-Preta program: The intervention for minors is delivered through an online platform, structured into 9 sessions of 45 minutes each, over 3 months. Weekly, platform-guided activities are proposed for classroom use with minimal teacher interaction, along with voluntary at-home activities.
  Other Names: PRETA Program
  Arms: Intervention Group

SUMMARY:
Background:

Eating Disorders (ED) are mental health conditions, characterized by pathological behaviors toward food intake or a persistent obsession with weight control. EDs have a high prevalence among pre-adolescents in developed countries and pose a significant economic burden. Preventive interventions targeting at-risk populations for ED have proven effective. The use of Information and Communication Technologies (ICTs) facilitates access to larger population groups while also reducing costs.

Objectives:

* Develop and validate a universally applied intervention (PRETA), mediated by ICTs, to reduce eating-disorder risk and modifiable risk factors, through cultural adaptation and adjustment of the POtsdam Prevention at Schools (POPS) Program to preadolescents.
* Assess the efficacy of the PRETA Program through a randomized controlled trial (RCT).
* Evaluate the efficiency of the PRETA Program from a social perspective. Methodology The PRETA Program uses 9 online sessions with interactive activities for pre- adolescents, plus education for their families and teachers.

Its content includes addressing key factors in the development of ED, such as eating habits, beauty standards, and media literacy, as well as activities aimed at strengthening psychological dimensions (self-esteem, emotional regulation, problem-solving, psychological flexibility, and resilience) and social skills, including communication styles and distinguishing between jokes and bullying.

The study involves schools being randomly assigned to either the PRETA Program or regular health activities. The effect of the intervention will be evaluated 3 months after its start.

DETAILED DESCRIPTION:
A matched-pair cluster random allocation will be used, with schools being asigned as clusters. Six schools will be assigned to each group.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the fifth or sixth year of primary education.
* Informed consent provided by the student's legal guardians and responsible teacher to participate.

Exclusion Criteria:

* Significant comprehension difficulties that limit adequate participation in the program and questionnaires.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1068 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Children's Eating Attitudes Test (ChEAT-26) Questionnaire score | Before and inmediately after the intervention
  The ChEAT is an adaptation of the EAT-26 for children is a 26 items scored on a 6-option Likert scale. It is a validated, self-administered questionnaire in Spanish for children aged 8 and older, with a reading level of 5th grade. The questionnaire focuses on identifying issues related to a persistent concern with food, eating patterns, and abnormal attitudes for this age group. The total score is obtained by summing all items, resulting in a range from 0 to 78 points. A total score above 20 points may indicate a possible presence of ED

SECONDARY OUTCOMES:
Evaluation of body image measured with the Adapted Contour Drawing Rating Scale (A-CDRS) visual analog scale. | Before and inmediately after the intervention
  It consists of 9 male and 9 female figure outlines that increase in size as the score increases. This scale measures the level of satisfaction with one's own body image. The degree of satisfaction or discrepancy index is obtained by calculating the difference between the desired and perceived images. A difference of 2 points is associated with body image disturbance. Age-appropriate images adapted for children aged 10 to 13 years will be used.
Body dissatisfaction, bulimia, and drive for thinness measured with the Spanish version of the Eating Disorder Inventory-2 (EDI-2). | Before and inmediately after the intervention
  The Eating Disorders Inventory-2 is a self-report instrument consisting of 91 items assessing psychological and behavioral traits associated with eating disorders, primarily anorexia and bulimia nervosa, across 11 different subscales. The response scale is a six-point Likert scale ranging from 0 (never) to 5 (always). The total score is obtained by summing all responses; a higher score indicates a greater presence of the trait.
Internalization of the current aesthetic model and media pressure using the Spanish version of the Sociocultural Attitudes Towards Appearance Questionnaire-4 | Before and inmediately after the intervention
  The original instrument includes 5 subscales; however, in this study, only the subscales related to body image internalization will be applied: the current aesthetic model based on thinness and the current aesthetic model based on athletic build (10 items), and the pressure to meet beauty ideals promoted by the media (4 items). Items are answered on a 5-point Likert scale, ranging from 1 "completely disagree" to 5 "completely agree." The score is calculated by summing all items; a higher score indicates greater internalization and influence of the aesthetic body model.
Evaluation of global self-esteem measured with the Rosenberg Self-Esteem Scale | Before and inmediately after treatment
  consists of 10 items that assess global self-esteem in adolescents, including elements focused on feelings of self-respect and self-acceptance. The first 5 items are positively worded and scored from 4 (strongly agree) to 1 (strongly disagree); the last 5 items are negatively worded and scored from 1 (strongly agree) to 4 (strongly disagree). The total score is obtained by summing all item responses. A score above 30 indicates high self-esteem, a score between 26 and 29 is considered medium self-esteem, and a score below 25 reflects low self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Ramallo-Fariña, PhD in Biomedical Sciences, Principal Investigator — Servicio de Evaluación del Servicio Canario de la Salud
Locations (1):
- Servicio de Evaluación y Planificación del Servicio Canario de Salud, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request. The data to be shared will include all IPD that underlie results in a publication, as well as the statistical analysis plan, informed consent form and the analytic code.
  All sensitive data will be anonymized to ensure the privacy and confidentiality of the participants.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All IPD, except for data related to outcome measures obtained at the post-intervention stage, will be available for sharing prior to the study's completion. The complete IPD will be available for sharing six months after the study's conclusion.
Access Criteria: As an access criterion for Individual Participant Data (IPD), it is required that no information be requested that could compromise the anonymity of participants. This ensures adherence to ethical research standards and the protection of personal data, safeguarding the confidentiality and privacy of all individuals involved.

REFERENCES:
- [Derived] Ramallo-Farina Y, Del Pino-Sedeno T, Pinto Robayna B, Capafons-Sosa JI, Cuesta-Rubio M, Garcia-Bello MA, Torres-Castano A, Vallejo Torres L, Benitez Brito N, Martin Corral J, Hernandez Rodriguez AI, Diaz Melian CD, Paz Lopez M, Gonzalez-Gonzalez CS. Effectiveness and cost-effectiveness of an online school-based programme to reduce eating disorder risk factors in preadolescents (PRETA): protocol for a cluster-randomised controlled trial. BMJ Open. 2025 Oct 14;15(10):e104014. doi: 10.1136/bmjopen-2025-104014. PMID 41087111